CLINICAL TRIAL: NCT00286494
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of SYR110322 (SYR-322) When Used in Combination With Pioglitazone in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study of Alogliptin Combined With Pioglitazone in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322-TZD-009; 2005-004669-40 (EudraCT Number); U1111-1113-8552 (Registry Identifier: WHO)
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Active Comparator)
  Interventions: Drug: Pioglitazone
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin and pioglitazone
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin and pioglitazone

INTERVENTIONS:
Drug: Alogliptin and pioglitazone — Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 30 mg or 45 mg, tablets, orally, once daily for up to 26 weeks
  Other Names: SYR110322; Alogliptin; AD-4833; Pioglitazone; Actos; SYR-322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin and pioglitazone — Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 30 mg or 45 mg, tablets, orally, once daily for up to 26 weeks
  Other Names: SYR110322; Alogliptin; AD-4833; Pioglitazone; Actos; SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Pioglitazone — Alogliptin placebo-matching tablets, orally, once daily and pioglitazone 30 mg or 45 mg, tablets, orally, once daily for up to 26 weeks
  Other Names: AD-4833; Actos
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of alogliptin, once daily (QD), combined with pioglitazone in adults with type 2 diabetes mellitus

DETAILED DESCRIPTION:
There are approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, of which 90% to 95% are type 2. The prevalence of type 2 diabetes varies among racial and ethnic populations and has been shown to correlate with age, obesity, family history, history of gestational diabetes, and physical inactivity. Over the next decade, a marked increase in the number of adults with diabetes mellitus is expected.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of dipeptidyl peptidase IV will improve glycemic (glucose) control in patients with type 2 diabetes.

The aim of the current study is to evaluate the efficacy of alogliptin in combination with pioglitazone in subjects who are inadequately controlled on a thiazolidinedione (pioglitazone or rosiglitazone) alone or in combination with metformin or a sulfonylurea. Individuals who participate in this study will be required to commit to a screening visit and up to 14 additional visits at the study center. Study participation is anticipated to be about 34 weeks (or 8.5 months).

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of type 2 diabetes mellitus currently treated with a thiazolidinedione either alone or in combination with metformin or a sulfonylurea but who are experiencing inadequate glycemic control. The subject should have received the thiazolidinedione therapy (rosiglitazone or pioglitazone) either alone or in combination with metformin or a sulfonylurea for at least the 3 months prior to Screening and must have been on a stable dose for all their antidiabetic treatments for at least the month prior to Screening.
* No treatment with antidiabetic agents other than a thiazolidinedione alone or in combination with either metformin or a sulfonylurea within the 3 months prior to Screening. (Exception: if a subject has received other antidiabetic therapy for less than 7 days within the 3 months prior to Screening.)
* Body mass index greater than or equal to 23 kg/m2 and less than or equal to 45 kg/m2
* Fasting C-peptide concentration greater than or equal to 0.8 ng per mL. (If this screening criterion is not met, the subject still qualifies if C-peptide is greater than or equal to 1.5 ng per mL after a challenge test.)
* Glycosylated hemoglobin concentration between 7.0% and 10.0%, inclusive.
* If regular use of other, non-excluded medications, must be on a stable dose for at least the 4 weeks prior to Screening. However, as needed use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
* Systolic blood pressure less than or equal to 180 mm Hg and diastolic pressure less than or equal to 110 mm Hg.
* Hemoglobin greater than or equal to 12 g per dL for males and greater than or equal to10 g per dL for females.
* Alanine aminotransferase less than or equal to 2.5 times the upper limit of normal.
* Serum creatinine less than or equal to 2.0 mg per dL.
* Thyroid-stimulating hormone level less than or equal to the upper limit of the normal range and the subject is clinically euthyroid.
* Neither pregnant nor lactating.
* Female subjects of childbearing potential must be practicing adequate contraception. Adequate contraception must be practiced for the duration of participation in the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibits the subject from completing the study.
* Able and willing to provide written informed consent.

Exclusion Criteria

* Urine albumin to creatinine ratio of greater than 1000 μg per mg at Screening. If elevated, the subject may be rescreened within 1 week.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening. (A history of treated cervical intraepithelial neoplasia I or cervical intraepithelial neoplasia II is allowed.)
* History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* History of treated diabetic gastric paresis.
* New York Heart Association Class III or IV heart failure regardless of therapy. Currently treated subjects who are stable at Class I or II are candidates for the study.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* History of a psychiatric disorder that will affect the subject's ability to participate in the study.
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors.
* History of alcohol or substance abuse within the 2 years prior to Screening.
* Receipt of any investigational drug within the 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within the 3 months prior to Screening.
* Prior treatment in an investigational study of alogliptin.
* Excluded Medications:

  * Treatment with antidiabetic agents other than a thiazolidinedione alone or in combination with either metformin or a sulfonylurea is not allowed within the 3 months prior to Screening and through the completion of the end-of-treatment/early termination procedures.
  * Treatment with weight-loss drugs, any investigational antidiabetics, or oral or systemically injected glucocorticoids is not allowed from 3 months prior to randomization through the completion of the end-of-treatment/early termination procedures. Inhaled corticosteroids are allowed.

Subjects must not take any medications, including over-the-counter products, without first consulting with the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (77):
- United States (64):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - Artesia, California
  - Fresno, California
  - Mission Viejo, California
  - Northridge, California
  - Orange, California
  - San Diego, California
  - Walnut Creek, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Cocoa Beach, Florida
  - Hollywood, Florida
  - Kissimmee, Florida
  - Longwood, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Saint Cloud, Florida
  - Tampa, Florida
  - Lawrenceville, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Avon, Indiana
  - Elkhart, Indiana
  - Evansville, Indiana
  - Lafayette, Indiana
  - Erlanger, Kentucky
  - Baltimore, Maryland
  - Sudbury, Massachusetts
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Pinehurst, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Lansdale, Pennsylvania
  - West Grove, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Cookeville, Tennessee
  - Milan, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Texarkana, Texas
  - Burlington, Vermont
- Multiple Cities, Argentina
- Multiple Cities, Australia
- Multiple Cities, Brazil
- Multiple Cities, Czechia
- Multiple Cities, Germany
- Multiple Cities, Guatemala
- Multiple Cities, Hungary
- Multiple Cities, India
- Multiple Cities, Mexico
- Multiple Cities, Netherlands
- Multiple Cities, New Zealand
- Multiple Cities, Peru
- Multiple Cities, South Africa

REFERENCES:
- [Result] Pratley RE, Reusch JE, Fleck PR, Wilson CA, Mekki Q; Alogliptin Study 009 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor alogliptin added to pioglitazone in patients with type 2 diabetes: a randomized, double-blind, placebo-controlled study. Curr Med Res Opin. 2009 Oct;25(10):2361-71. doi: 10.1185/03007990903156111. PMID 19650752
- [Result] Pratley RE, McCall T, Fleck PR, Wilson CA, Mekki Q. Alogliptin use in elderly people: a pooled analysis from phase 2 and 3 studies. J Am Geriatr Soc. 2009 Nov;57(11):2011-9. doi: 10.1111/j.1532-5415.2009.02484.x. Epub 2009 Sep 30. PMID 19793357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 125 investigative sites in 13 countries from 24 February 2006 to 02 August 2007.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled in one of 3, once-daily (QD) treatment groups.
Groups:
- Placebo: Alogliptin placebo-matching tablets, orally, once daily and pioglitazone 30 mg or 45 mg, tablets, orally, once daily for up to 26 weeks.
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 30 mg or 45 mg, tablets, orally, once daily for up to 26 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 30 mg or 45 mg, tablets, orally, once daily for up to 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Started | 97 | 197 | 199
Completed | 71 | 153 | 160
Not Completed | 26 | 44 | 39
Not completed — Hyperglycemic rescue | 12 | 19 | 18
Not completed — Withdrawal by Subject | 2 | 10 | 9
Not completed — Adverse Event | 3 | 8 | 6
Not completed — Physician Decision | 5 | 5 | 1
Not completed — Lost to Follow-up | 3 | 1 | 3
Not completed — Protocol Violation | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Total
Number analyzed (Participants) | 97 | 197 | 199 | 493
Age, Customized [Number; unit: participants]
  <65 years | 83 | 165 | 160 | 408
  Between 65 and 74 years | 10 | 29 | 34 | 73
  ≥75 years | 4 | 3 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 88 | 74 | 206
  Male | 53 | 109 | 125 | 287

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26.
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 26 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 196 | 195
percentage of Glycosylated Hemoglobin | -0.19 (0.081) | -0.66 (0.056) | -0.80 (0.056)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Null Hypothesis: No difference between treatment and placebo arms in change from baseline in glycosylated hemoglobin at wk 26. Sample size calculated based on normally distributed means. For comparison of either dose vs. placebo (2-sample t-test), study sample size >=500 subjects had 95% power to detect a treatment difference as small as 0.4% in the supportive per protocol analysis set assuming SD=0.8%, 2-sided >0.05 significance level and >=80% of subjects meeting per protocol criteria; Test type: Superiority or Other; p < 0.001, ANCOVA — A step-down strategy was used for the primary analysis. First, the 25mg dose was compared to placebo at the 2-sided 0.05 significance level. The 12.5 mg dose was compared to placebo only if the comparison of the 25mg dose to placebo was significant; Treatment, treatment regimen and geographic region as class variables; baseline pioglitazone dose and baseline value for the endpoint as covariates; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.67 to -0.28] — Negative mean treatment difference indicates larger decrease from baseline (more negative change from baseline) in the alogliptin arm compared to the placebo arm
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.80 to -0.41] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF).). Smaller "n" at earlier timepoints due to unavailable prior values to carry forward.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 90 | 182 | 176
percentage of Glycosylated Hemoglobin | -0.14 (0.042) | -0.40 (0.029) | -0.45 (0.030)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment, geographic region and baseline treatment regimen as class variables; baseline pioglitazone dose and value for endpoint as covariates; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.36 to -0.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.41 to -0.21] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 196 | 195
percentage of Glycosylated Hemoglobin | -0.18 (0.061) | -0.60 (0.042) | -0.73 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.56 to -0.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.69 to -0.40] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 196 | 195
percentage of Glycosylated Hemoglobin | -0.23 (0.069) | -0.70 (0.048) | -0.82 (0.048)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.63 to -0.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.75 to -0.43] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 196 | 195
percentage of Glycosylated Hemoglobin | -0.26 (0.076) | -0.70 (0.053) | -0.84 (0.053)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.63 to -0.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.76 to -0.40] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 196 | 195
percentage of Glycosylated Hemoglobin | -0.27 (0.078) | -0.68 (0.055) | -0.82 (0.055)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.60 to -0.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.74 to -0.36] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 1).
Description: The change between the value of fasting plasma glucose collected at final visit or week 1 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 1.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF).Smaller "n" at earlier timepoints due to unavailable prior values to carry forward.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 88 | 176 | 171
mg/dL | -2.7 (3.11) | -14.2 (2.20) | -18.2 (2.22)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -11.4, 95% CI 2-sided [-18.9 to -3.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -15.5, 95% CI 2-sided [-23.0 to -8.0] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 189 | 193
mg/dL | -1.8 (2.97) | -21.0 (2.13) | -21.2 (2.10)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -19.2, 95% CI 2-sided [-26.4 to -11.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -19.4, 95% CI 2-sided [-26.6 to -12.3] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 194 | 197
mg/dL | -3.1 (2.88) | -23.7 (2.04) | -26.0 (2.02)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -20.6, 95% CI 2-sided [-27.5 to -13.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -23.0, 95% CI 2-sided [-29.9 to -16.0] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 196 | 197
mg/dL | -6.1 (3.26) | -22.6 (2.30) | -27.1 (2.29)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -16.5, 95% CI 2-sided [-24.4 to -8.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -21.1, 95% CI 2-sided [-28.9 to -13.3] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 196 | 197
mg/dL | -9.9 (3.33) | -20.4 (2.34) | -26.2 (2.33)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.011, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-18.5 to -2.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -16.3, 95% CI 2-sided [-24.3 to -8.3] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 16).
Description: The change between the value of fasting plasma glucose collected at week 16 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 196 | 197
mg/dL | -8.3 (3.71) | -18.3 (2.61) | -22.8 (2.60)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.029, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-18.9 to -1.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -14.4, 95% CI 2-sided [-23.3 to -5.5] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 20).
Description: The change between the value of fasting plasma glucose collected at week 20 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 196 | 197
mg/dL | -6.4 (3.58) | -21.9 (2.52) | -21.6 (2.51)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -15.6, 95% CI 2-sided [-24.2 to -6.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -15.2, 95% CI 2-sided [-23.8 to -6.7] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 26).
Description: The change between the value of fasting plasma glucose collected at week 26 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 196 | 197
mg/dL | -5.7 (3.81) | -19.7 (2.68) | -19.9 (2.67)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -13.9, 95% CI 2-sided [-23.1 to -4.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -14.1, 95% CI 2-sided [-23.3 to -5.0] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Number of Participants With Marked Hyperglycemia (Fasting Plasma Glucose ≥ 200 mg Per dL).
Description: The number of participants with a fasting plasma glucose value greater than or equal to 200 mg per dL during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set) and had at least 1 post-baseline FPG measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 196 | 198
participants | 43 | 49 | 43
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline pioglitazone dose, baseline treatment regimen, & baseline HbA1c; Odds Ratio (OR) = 0.271, 95% CI 2-sided [0.147 to 0.499] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 0.235, 95% CI 2-sided [0.126 to 0.438] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

16. Secondary Outcome: Number of Participants Requiring Rescue.
Description: The number of participants requiring rescue for failing to achieve pre-specified glycemic targets during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set)and at least 1 post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 196 | 199
participants | 12 | 19 | 18
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.266, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline pioglitazone dose, baseline treatment regimen & baseline HbA1c; Odds Ratio (OR) = 0.628, 95% CI 2-sided [0.277 to 1.425] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.315, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 0.658, 95% CI 2-sided [0.292 to 1.487] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

17. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 4).
Description: The change between the value of fasting proinsulin collected at week 4 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF). Smaller "n" at earlier timepoints due to unavailable prior values to carry forward.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 87 | 172 | 169
pmol/L | -0.7 (1.74) | -7.0 (1.24) | -5.6 (1.25)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-10.6 to -2.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.023, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-9.1 to -0.7] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 8).
Description: The change between the value of fasting proinsulin collected at week 8 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 92 | 186 | 188
pmol/L | -2.3 (1.70) | -6.5 (1.19) | -3.7 (1.19)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.043, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-8.3 to -0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.489, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.5 to 2.6] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 12).
Description: The change between the value of fasting proinsulin collected at week 12 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 92 | 186 | 188
pmol/L | 0.6 (1.88) | -3.6 (1.33) | -3.8 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.068, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-8.8 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.056, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-8.9 to 0.1] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 16).
Description: The change between the value of fasting proinsulin collected at week 16 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 92 | 186 | 188
pmol/L | -3.1 (1.89) | -3.5 (1.33) | -3.1 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.884, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-4.9 to 4.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.993, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-4.5 to 4.5] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 20).
Description: The change between the value of fasting proinsulin collected at week 20 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 92 | 186 | 188
pmol/L | -0.9 (1.67) | -6.2 (1.18) | -3.9 (1.17)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.009, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-9.4 to -1.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.143, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-7.0 to 1.0] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 26).
Description: The change between the value of fasting proinsulin collected at week 26 or final visit and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 92 | 186 | 188
pmol/L | -1.0 (1.9) | -5.1 (1.34) | -1.7 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.080, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-8.6 to 0.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.782, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-5.2 to 3.9] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Change From Baseline in Insulin (Week 4).
Description: The change between the value of insulin collected at week 4 and insulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 86 | 166 | 165
mcIU/mL | -0.09 (0.694) | -1.08 (0.501) | -0.97 (0.501)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.249, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-2.68 to 0.70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.303, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-2.56 to 0.80] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Change From Baseline in Insulin (Week 8).
Description: The change between the value of insulin collected at week 8 and insulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
mcIU/mL | -0.17 (0.748) | -0.82 (0.531) | 0.21 (0.522)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.478, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-2.46 to 1.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.674, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-1.41 to 2.17] — [estimate comment as in outcome 1, analysis 1]

25. Secondary Outcome: Change From Baseline in Insulin (Week 12).
Description: The change between the value of insulin collected at week 12 and insulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
mcIU/mL | 0.00 (1.085) | 0.43 (0.771) | -0.58 (0.757)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.743, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-2.18 to 3.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.662, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-3.18 to 2.02] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Change From Baseline in Insulin (Week 16).
Description: The change between the value of insulin collected at week 16 and insulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
mcIU/mL | -0.85 (0.701) | -0.10 (0.501) | -0.16 (0.492)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.390, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.75, 95% CI 2-sided [-0.96 to 2.45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.423, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-1.00 to 2.38] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Change From Baseline in Insulin (Week 20).
Description: The change between the value of insulin collected at week 20 and insulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
mcIU/mL | -0.19 (0.690) | -0.40 (0.490) | -0.33 (0.481)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.807, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.87 to 1.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.867, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-1.79 to 1.51] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Change From Baseline in Insulin (Week 26).
Description: The change between the value of insulin collected at week 26 and insulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
mcIU/mL | -0.81 (0.711) | -0.19 (0.505) | 0.00 (0.495)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.483, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-1.10 to 2.33] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.352, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-0.89 to 2.51] — [estimate comment as in outcome 1, analysis 1]

29. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 4).
Description: The change between the ratio value of proinsulin and insulin collected at week 4 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 86 | 166 | 165
ratio | 0.006 (0.0144) | -0.051 (0.0104) | -0.053 (0.0104)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.057, 95% CI 2-sided [-0.092 to -0.022] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.059, 95% CI 2-sided [-0.093 to -0.024] — [estimate comment as in outcome 1, analysis 1]

30. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 8).
Description: The change between the ratio value of proinsulin and insulin collected at week 8 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
ratio | -0.006 (0.0145) | -0.055 (0.0103) | -0.057 (0.0101)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.006, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.084 to -0.014] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.004, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.086 to -0.016] — [estimate comment as in outcome 1, analysis 1]

31. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 12).
Description: The change between the ratio value of proinsulin and insulin collected at week 12 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
ratio | 0.017 (0.0190) | -0.029 (0.0135) | -0.040 (0.0132)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.050, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.046, 95% CI 2-sided [-0.092 to 0.000] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.014, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.057, 95% CI 2-sided [-0.102 to -0.012] — [estimate comment as in outcome 1, analysis 1]

32. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 16).
Description: The change between the ratio value of proinsulin and insulin collected at week 16 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
ratio | -0.015 (0.0153) | -0.042 (0.0109) | -0.045 (0.0107)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.144, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.027, 95% CI 2-sided [-0.064 to 0.009] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.105, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.030, 95% CI 2-sided [-0.067 to 0.006] — [estimate comment as in outcome 1, analysis 1]

33. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 20).
Description: The change between the ratio value of proinsulin and insulin collected at week 20 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
ratio | 0.012 (0.0168) | -0.047 (0.0119) | -0.040 (0.0117)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.004, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.059, 95% CI 2-sided [-0.100 to -0.019] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.012, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.092 to -0.011] — [estimate comment as in outcome 1, analysis 1]

34. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 26).
Description: The change between the ratio value of proinsulin and insulin collected at week 26 or final visit and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 91 | 181 | 187
ratio | 0.015 (0.0185) | -0.035 (0.0131) | -0.022 (0.0129)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.028, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.050, 95% CI 2-sided [-0.095 to -0.005] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.093, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.038, 95% CI 2-sided [-0.082 to 0.006] — [estimate comment as in outcome 1, analysis 1]

35. Secondary Outcome: Change From Baseline in C-peptide (Week 4).
Description: The change between the value of C-peptide collected at week 4 and C-peptide collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 90 | 181 | 175
ng/mL | -0.144 (0.1108) | -0.156 (0.0783) | -0.088 (0.0794)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.928, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.280 to 0.255] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.683, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.056, 95% CI 2-sided [-0.212 to 0.324] — [estimate comment as in outcome 1, analysis 1]

36. Secondary Outcome: Change From Baseline in C-peptide (Week 8).
Description: The change between the value of C-peptide collected at week 8 and C-peptide collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 195 | 194
ng/mL | -0.111 (0.1127) | -0.117 (0.0787) | 0.023 (0.0788)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.967, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.277 to 0.265] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.327, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.135, 95% CI 2-sided [-0.135 to 0.405] — [estimate comment as in outcome 1, analysis 1]

37. Secondary Outcome: Change From Baseline in C-peptide (Week 12).
Description: The change between the value of C-peptide collected at week 12 and C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 195 | 194
ng/mL | -0.017 (0.1226) | -0.085 (0.0856) | -0.067 (0.0856)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.649, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.068, 95% CI 2-sided [-0.363 to 0.226] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.735, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.344 to 0.243] — [estimate comment as in outcome 1, analysis 1]

38. Secondary Outcome: Change From Baseline in C-peptide (Week 16).
Description: The change between the value of C-peptide collected at week 16 and C-peptide collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 195 | 194
ng/mL | -0.290 (0.1135) | -0.071 (0.0793) | -0.052 (0.0793)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.114, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.220, 95% CI 2-sided [-0.053 to 0.492] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.086, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.238, 95% CI 2-sided [-0.033 to 0.510] — [estimate comment as in outcome 1, analysis 1]

39. Secondary Outcome: Change From Baseline in C-peptide (Week 20).
Description: The change between the value of C-peptide collected at week 20 and C-peptide collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 195 | 194
ng/mL | -0.255 (0.1029) | -0.228 (0.0718) | -0.123 (0.0719)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.835, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.221 to 0.273] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.296, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [-0.115 to 0.378] — [estimate comment as in outcome 1, analysis 1]

40. Secondary Outcome: Change From Baseline in C-peptide (Week 26).
Description: The change between the value of C-peptide collected at week 26 or final visit and C-peptide collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 95 | 195 | 194
ng/mL | -0.356 (0.1071) | -0.233 (0.0748) | -0.133 (0.0748)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.349, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.123, 95% CI 2-sided [-0.134 to 0.380] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.089, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.223, 95% CI 2-sided [-0.034 to 0.479] — [estimate comment as in outcome 1, analysis 1]

41. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 6.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 6.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 197 | 199
participants | 5 | 34 | 41
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.003, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 4.815, 95% CI 2-sided [1.736 to 13.358] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 5.533, 95% CI 2-sided [2.017 to 15.176] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

42. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.0%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin less (the percentage of hemoglobin that is bound to glucose) than or equal to 7.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 197 | 199
participants | 33 | 87 | 98
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.029, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 1.903, 95% CI 2-sided [1.067 to 3.393] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, baseline pioglitazone dose, baseline treatment regiment & baseline HbA1c; Odds Ratio (OR) = 2.301, 95% CI 2-sided [1.291 to 4.100] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

43. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 7.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 197 | 199
participants | 47 | 127 | 141
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 2.783, 95% CI 2-sided [1.547 to 5.005] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 3.917, 95% CI 2-sided [2.147 to 7.146] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

44. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 0.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 0.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 197 | 199
participants | 26 | 118 | 128
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 4.134, 95% CI 2-sided [2.392 to 7.146] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 5.247, 95% CI 2-sided [3.027 to 9.094] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

45. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 197 | 199
participants | 12 | 64 | 73
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 3.670, 95% CI 2-sided [1.789 to 7.532] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 4.693, 95% CI 2-sided [2.303 to 9.560] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

46. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 197 | 199
participants | 5 | 32 | 37
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.015, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 3.800, 95% CI 2-sided [1.300 to 11.107] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.002, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 5.196, 95% CI 2-sided [1.806 to 14.950] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

47. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 2.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 2.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 97 | 197 | 199
participants | 3 | 12 | 14
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.364, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 1.959, 95% CI 2-sided [0.459 to 8.362] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.146, Regression, Logistic; [statistical method as in outcome 16, analysis 1]; Odds Ratio (OR) = 2.849, 95% CI 2-sided [0.696 to 11.672] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

48. Secondary Outcome: Change From Baseline in Body Weight (Week 8).
Description: The change between Body Weight measured at week 8 and Body Weight measured at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 93 | 190 | 186
kg | 0.36 (0.228) | 0.46 (0.160) | 0.39 (0.161)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.718, ANCOVA — No multiplicity adjustments; Treatment, geographic region and baseline treatment regimen as class variables; baseline pioglitazone dose,baseline value for endpoint as covariates; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.45 to 0.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.906, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.52 to 0.58] — [estimate comment as in outcome 1, analysis 1]

49. Secondary Outcome: Change From Baseline in Body Weight (Week 12).
Description: The change between Body Weight measured at week 12 and Body Weight measured at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 94 | 193 | 189
kg | 0.60 (0.267) | 0.74 (0.187) | 0.64 (0.188)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.672, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.50 to 0.78] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.922, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.61 to 0.67] — [estimate comment as in outcome 1, analysis 1]

50. Secondary Outcome: Change From Baseline in Body Weight (Week 20).
Description: The change between Body Weight measured at week 20 and Body Weight measured at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 94 | 193 | 189
kg | 0.94 (0.318) | 1.14 (0.222) | 0.93 (0.224)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.607, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.56 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.985, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.77 to 0.76] — [estimate comment as in outcome 1, analysis 1]

51. Secondary Outcome: Change From Baseline in Body Weight (Week 26).
Description: The change between Body Weight measured at week 26 or final visit and Body Weight measured at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 94 | 193 | 189
kg | 1.04 (0.329) | 1.46 (0.230) | 1.09 (0.232)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.294, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.37 to 1.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.900, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.74 to 0.84] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious event) after the last dose of double-blind drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Serious Adverse Events (participants affected / at risk) | 4/97 | 5/198 | 13/199
Other Adverse Events (participants affected / at risk) | 38/97 | 76/198 | 79/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | Alogliptin 12.5 mg QD (N=198) | Alogliptin 25 mg QD (N=199)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | Alogliptin 12.5 mg QD (N=198) | Alogliptin 25 mg QD (N=199)
Oedema peripheral (General disorders) | 7 | 12 | 11
Nasopharyngitis (Infections and infestations) | 6 | 8 | 14
Sinusitis (Infections and infestations) | 6 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 11 | 10
Influenza (Infections and infestations) | 4 | 3 | 11
Bronchitis (Infections and infestations) | 5 | 4 | 3
Headache (Nervous system disorders) | 4 | 8 | 10
Nausea (Gastrointestinal disorders) | 2 | 9 | 6
Urinary tract infection (Infections and infestations) | 1 | 9 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 8
Hypertension (Vascular disorders) | 2 | 6 | 8
Dizziness (Nervous system disorders) | 2 | 7 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Fatigue (General disorders) | 3 | 4 | 4
Joint injury (Injury, poisoning and procedural complications) | 3 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.